CLINICAL TRIAL: NCT00079131
Title: A Phase II Study of G3139 (Genasense ™) in Patients With Merkel Cell Carcinoma
Brief Title: Oblimersen in Treating Patients With Merkel Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01446; 03-105; CDR0000354418; NCI-5907; MSKCC-03105; N01CM62207 (NIH); N01CM62206 (NIH)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Recurrent Neuroendocrine Carcinoma of the Skin; Stage I Neuroendocrine Carcinoma of the Skin; Stage II Neuroendocrine Carcinoma of the Skin; Stage III Neuroendocrine Carcinoma of the Skin; Stage IV Neuroendocrine Carcinoma of the Skin
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — oblimersen

ARMS (1):
- Treatment (oblimersen sodium) (Experimental): Patients receive oblimersen IV continuously on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: oblimersen sodium; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: oblimersen sodium — Given IV
  Other Names: augmerosen; G3139; G3139 bcl-2 antisense oligodeoxynucleotide; Genasense
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well oblimersen works in treating patients with Merkel cell cancer. Biological therapies, such as oblimersen, may interfere with the growth of tumor cells and slow the growth of Merkel cell carcinoma (skin cancer).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall response rate in patients with Merkel cell carcinoma treated with oblimersen.

SECONDARY OBJECTIVES:

I. Determine the time to progression in patients treated with this drug. II. Determine the response duration in patients treated with this drug. III. Determine the safety and tolerability of this drug in these patients. IV. Determine the pharmacodynamic effects of this drug on bcl-2 expression and apoptosis in tumor biopsy specimens from these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oblimersen IV continuously on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Merkel cell carcinoma

  * Metastatic OR regionally recurrent disease
  * Localized disease not amenable to curative therapy (surgery or radiotherapy) also allowed
* Measurable disease

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No known brain metastases

  * Previously resected or irradiated brain metastases allowed if stable for at least the past 3 months and no evidence of neurological compromise exists
* Performance status - Karnofsky 60-100%
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* WBC >= 3,000/mm^3
* AST/ALT =< 2.5 times upper limit of normal
* Bilirubin normal
* INR =< 1.5
* Creatinine normal
* Creatinine clearance >= 60 mL/min
* No atrial fibrillation unless stable for at least the past 6 months
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Adequate venous access
* No peripheral neuropathy > grade 1
* No active or ongoing infection
* No other concurrent uncontrolled illness
* No prior grade 3 or 4 anaphylactic reaction to phosphorothioate oligonucleotide
* No psychiatric illness or social situation that would preclude study compliance
* More than 3 weeks since prior chemotherapy and recovered
* More than 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to 25% or more of bone marrow
* More than 3 weeks since prior investigational therapy and recovered
* No prior oblimersen
* No other concurrent investigational agents
* No concurrent anticoagulation except 1 mg of warfarin for mediport patency
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2004-01; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 3 years

SECONDARY OUTCOMES:
Time to progression | Interval between the start of treatment and until the criteria for progression are met, assessed up to 3 years
  Progression-free survival probabilities will be computed using Kaplan-Meier methods.
Occurrence of adverse events, assessed using revised NCI CTC version 3.0 | Within 30 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ki Chung, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States